CLINICAL TRIAL: NCT04929340
Title: Prevention of Recurrent Childhood Caries With Probiotic Supplement, a Randomized Controlled Trial
Brief Title: Prevention of Recurrent Caries With Lactobacilli PRECAL
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment on hold since spring 2020 due to Covid-19 pandemic
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Pamela Hasselof, Principal Investigator, senior consultant dentist, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OD5.1-8-17
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Dental Caries in Children
Keywords: Early childhood caries; Probiotic bacteria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: yellow / blue dots on the bottles indicates different groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): 5 drops each day before bedtime but after toothbrushing. L. reuteri DSM 17938, L. reuteri ATCC PTA 5289, with a minimum of 100 million live bacteria of each strain.
  Interventions: Other: Probiotic bacteria
- placebo (Placebo Comparator): 5 drops each day before bedtime but after toothbrushing. The placebo drops had identical composition color and taste but no probiotic bacteria.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Probiotic bacteria — The children are randomly allocated to a test or a control group with aid of computer-generated numbers at the time of consent. After the treatment, children in the test group are given 5 drops per day containing probiotic bacteria (Lactobacillus reuteri Protectis DSM 17938, Biogaia AB, Sweden) before bedtime. One dose consists of a minimum of 100 million live bacteria. Children in control group are given 5 drops per day (containing no bacteria).
  Other Names: Experimental
  Arms: experimental
Other: Placebo — Children in control group are given 5 drops per day (containing no bacteria).
  Arms: placebo

SUMMARY:
The aim of this study was to compare the effect of drops containing probiotic bacteria (Lactobacillus reuteri 17938, Lactobacillus reuteri PTA 5289, Biogaia AB, Sweden) on the incidence of dental caries with placebo drops in preschool children undergoing comprehensive restorative treatment under general anesthesia or conscious sedation. The project will be conducted at three specialist centers (Umeå University, Umeå, Sweden, Maxillo-facial unit, Halmstad Hospital, Sweden; Eastman Institute, Stockholm, Sweden) and employ a randomized placebo-controlled design with two parallel arms. The study will be performed double-blind and neither the parents nor the clinicians will be aware of the content of the drops. The follow-up period is one year.

ELIGIBILITY:
Inclusion Criteria:

* Preschool children, 2-5 year of age
* with Early childhood caries (ECC) or
* severe Early childhood caries (S-ECC)
* scheduled for restorations and extractions under general anesthesia or any form of sedation
* The obligate requirement is that the child should be fully treated and managed with aspect to caries within a period of not more than two months.

Exclusion Criteria:

* medically comprised children
* children with severe cognitive problems or dysfunctional families
* families planning to relocate within the next year

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
dental caries | 6 months
  dental caries (International Caries Detection and Assesment System, ICDAS level)
dental caries | 12 months
  dental caries (International Caries Detection and Assesment System, ICDAS level)

SECONDARY OUTCOMES:
visible supra-gingival plaque | 6 months
  presence of visible supragingival plaque on buccal surfaces upper anterior teeth (yes/no)
visible supra-gingival plaque | 12 months
  presence of visible supragingival plaque on buccal surfaces upper anterior teeth (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Hasslöf, Principal Investigator — Umeå University
Locations (3):
- Sweden (3):
  - Barntandvården Halmstad, Halmstad
  - Eastmaninstitutet Pedodonti, Stockholm, Stockholm
  - Tandläkarhögskolan Umeå, Umeå

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasslof P, Granqvist L, Stecksen-Blicks C, Twetman S. Prevention of Recurrent Childhood Caries with Probiotic Supplements: A Randomized Controlled Trial with a 12-Month Follow-Up. Probiotics Antimicrob Proteins. 2022 Apr;14(2):384-390. doi: 10.1007/s12602-022-09913-9. Epub 2022 Jan 26. PMID 35083729